CLINICAL TRIAL: NCT02938182
Title: A Prospective Trial to Evaluate the Effectiveness of Clopidogrel to Relieve Migraine With Right-to-left Shunt
Brief Title: Migraine Prophylaxis With Clopidogrel Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRS-2016-019
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clopidogrel (Experimental): clopidogrel tablet 75mg daily for three months
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: clopidogrel — clopidogrel troche 75 mg daily for three months
  Other Names: plavix

SUMMARY:
The underlying mechanisms of association between the right-to-left shunts (RLS) and migraine may concern with platelet aggregation and paradoxical embolization. The aim of the study is to evaluate the prophylactic effectiveness of clopidogrel for migraineurs with RLS.

DETAILED DESCRIPTION:
Many studies have shown an increased prevalence of right-to-left shunts in migraineurs. The underlying mechanisms of association between the right-to-left shunts (RLS) and migraine may concern with platelet aggregation and paradoxical embolization. In the present study, migraineurs without taking prophylactic medicines regularly will be given only clopidogrel 75 mg daily for three months. Migraineurs who are unresponsive to at least two commonly applied preventive medications, clopidogrel 75 mg daily will be added to his/her existing prophylactic migraine regimen for three months. Patients will be followed up at the third month and the sixth month for headache frequency, attack duration of headache, migraine disability assessment scale（MIDAS）scores, headache impact test（HIT-6）scores and visual analogue scale（VAS）scores. Investigators will evaluate the changes of these measurements between baseline and the follow-up time. The aim of the study is to evaluate the prophylactic effectiveness of clopidogrel for migraineurs with RLS.

ELIGIBILITY:
Inclusion Criteria:

* migraine with or without aura diagnosed by a neurologist according to the criteria of the International Headache Society (3nd edition)
* experience a minimum of two migraine attacks per month in a 3-month baseline phase
* without regular use of prophylactic treatments or unresponsive to two and more commonly applied preventive medications
* the presence of RLS confirmed by contrast-enhanced transcranial Doppler
* no positive findings in cranial CT and MRI

Exclusion Criteria:

* other types of headaches
* systemic chronic diseases, cerebrovascular disease, abnormal platelet or liver function
* history of head injury
* other contraindications to clopidogrel treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-10; Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Attack Duration of Headache at three months, h | three months

SECONDARY OUTCOMES:
Change from Baseline Headache Frequency per Month at three months, time | three months
Change from Baseline Visual Analogue Scale at three months, scores | three months
Change from Baseline Migraine Disability Assessment Scale at three months, scores | three months
Change from Baseline Headache Impact Test at three months, scores | three months

CONTACTS AND LOCATIONS:
Overall Officials: Guogang Luo, doctor, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
The information of the patients need to keep confidential.